CLINICAL TRIAL: NCT01605409
Title: Emergency Cardiopulmonary Bypass After Cardiac Arrest With Ongoing Cardiopulmonary Resuscitation - a Pilot Randomized Trial
Brief Title: Emergency Cardiopulmonary Bypass for Cardiac Arrest
Acronym: ECPB4OHCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Andreas Schober, MD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KLI196
Record Dates: First submitted 2012-05-22; First posted 2012-05-24 (Estimated); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Cardiac Arrest
Keywords: Refractory cardiac arrest; Emergency cardiopulmonary bypass; Extracorporeal life support in cardiac arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard ACLS (Active Comparator): Patients in the standard ACLS group will be resuscitated until ROSC or termination of efforts. If ROSC is achieved they will be transported to the emergency department and treated according to ERC guidelines and GCP.
  Interventions: Procedure: Standard ACLS
- ECPB (Experimental): ACLS provided for 15 minutes by EMS personnel according to current guidelines of the ERC.
  CPR during transportation will be performed by EMS personnel according to ERC guidelines.
  At the ED cannulation will be performed percutaneously if feasible. The femoral artery will be cannulated with a 17-19 - Fr and the femoral vein will be cannulated simultaneously with heparin coated 19-25 - Fr catheter or a smart cannula. An antegrade 8 - Fr cannula will be placed to supply perfusion for the cannulated leg if feasible. The procedures will be performed ultrasound-guided and the size of the cannulae will be adapted according to vessel size. Correct placement of the venous cannulae will be verified via ultrasound. Cardiopulmonary bypass will be performed by using the Lifebridge(Sorin®) or the Cardiohelp(Maquet®) ECMO device, according to protocol.
  Interventions: Procedure: Emergency cardiopulmonary bypass under ongoing CPR; Procedure: Standard ACLS

INTERVENTIONS:
Procedure: Emergency cardiopulmonary bypass under ongoing CPR — Emergency cardiopulmonary bypass under ongoing CPR
  Emergency cardiopulmonary bypass (ECMO: lifebridge (Sorin®) or cardiohelp(Maquet®) will be initiated percutaneously ultrasound guided, during CPR efforts at the Emergency department.
  Cannulae and tubing in use will be heparin coated. ECMO flow will be set to 70ml/kgBW/min. Anticoagulation will achieved with unfractionated heparin and monitored using ACT.
  Arms: ECPB
Procedure: Standard ACLS — Standard ACLS Standard ACLS provided by EMS personnel according to current guidelines of the European resuscitation council.
  Transportation:
  Transport will be initiated as soon as the patient achieves ROSC in the field and transportation is feasible. All patients will be admitted to the ED at the Vienna general hospital.
  Standard Post resuscitation Management:
  After admission to the ED post resuscitation care and standardized intensive care treatment will be provided according to Utstein protocol and current standards for good clinical practice and according to ILCOR recommendations. A crossover to the ECPB group is possible, if indicated by good clinical practice. If so, it will be counted as treatment failure in the standard ACLS group.
  If no ROSC can be achieved and the patient dies in the field pathological results will be obtained if feasible.

SUMMARY:
Cardiac arrest ist associated with a very poor prognosis. Even though resuscitation algorithms and postcardiac arrest care have been improved there is an urgent need for measures leading to a higher survival rate.

Emergency cardiopulmonary bypass (ECPB - artificial heart and lung outside the patients body) is a method which has shown good results in case reports and animal studies for cardiac arrest care.

The study will be performed as comparison between the new treatment option of ECPB versus the standard of care treatment.

Aim of our study is to determine the feasibility of ECPB installed in an emergency department to improve the rate of patients restoration of spontaneous circulation.

DETAILED DESCRIPTION:
Background: Out of hospital cardiac arrest is associated with a poor prognosis. Overall survival varies between 3% and 16% respectively. Measures to improve the chance of survival are urgently needed. If return of spontaneous circulation under competent cardiopulmonary resuscitation (CPR) measures is not achieved within the first 25 minutes the chance of survival decreases even further. Emergency Cardiopulmonary Bypass (ECPB) would be such a treatment option for these heavily compromised patients, as it has shown considerably good results used as resuscitation device for cardiac arrest in animal studies.

Material and Methods: This study will be performed as single center (university hospital) randomized, controlled and prospective pilot study comprising a highly experienced emergency department treating about 200 to 300 cardiac arrest patients a year. Two groups will be analyzed, a 'Standard ACLS´ group and an 'ECPB´ group. Each group will comprise 20 patients. Eligible are adult patients with witnessed out of hospital cardiac arrest, with presumed cardiac cause and without return of spontaneous circulation after a minimum of 15 minutes of advanced cardiac life support.

Patients in the 'Standard ACLS´ group will be resuscitated until return of spontaneous circulation or termination of efforts. The 'ECPB´ group will receive ongoing cardiopulmonary resuscitation during transport to the emergency department where ECPB will be installed. Necessary diagnostic examinations and therapeutic interventions for both groups will be performed according to guidelines for post resuscitation care and good clinical practice.

Primary outcome measure is the rate of sustained restoration of spontaneous circulation according to Utstein criteria. Secondary outcome measures are 24 hours survival, survival to ICU discharge, survival to hospital discharge, rate of best neurological recovery (cerebral performance category score 1 or 2) within 6 months after cardiac arrest and modified Rankin score at 6 months after cardiac arrest.

Patients in the 'Standard ACLS´ group receive standard treatment without any potential additional risks. The 'ECPB´ group receives standard advanced cardiac life support as well and has the predicted advantage of the extracorporeal oxygenation at the emergency department and coronary intervention even before return of spontaneous circulation.

Aim of this study: To compare current standard therapy for patients after out of hospital cardiac arrest (cardiopulmonary resuscitation until return of spontaneous circulation or termination of efforts) with a new concept of transportation with ongoing cardiopulmonary reanimation and installation of ECPB at the Emergency Department to improve survival.

ELIGIBILITY:
Inclusion Criteria:

Patients with witnessed out-of-hospital cardiac arrest, with presumed cardiac cause, immediate initiation of bystander CPR and without return of spontaneous circulation after a minimum of 15 minutes of advanced cardiac life support are eligible. Patients who do achieve ROSC at first but suffer rearrest afterwards and do not achieve ROSC again after 15 minutes of advanced cardiac life support are considered eligible as well.

Exclusion Criteria:

* Patients younger than 18 years or older than 75 years
* Traumatic cardiac arrest
* Cardiac arrest due to exsanguination, strangulation, hanging or drowning
* Accidental hypothermia as a cause of cardiac arrest
* Women suffering life-threatening amniotic fluid embolism
* Cardiac arrest due to pulmonary artery embolism
* Cardiac arrest due to intoxication
* Cardiac arrest due to intracranial hemorrhage
* Other initial ECG-rhythm than ventricular fibrillation
* Known or clinically apparent pregnancy
* Patients with an Allow-natural-death- (AND) or Do-not-attempt-resuscitation (DNAR) order or patients with a terminal illness
* Patients who, for any reason, can not be transported with ongoing CPR
* Insufficient quality of bystander CPR (at the discretion of the emergency physician or EMT)*
* Estimated transportation time exceeding 30 minutes
* Patients with psychiatric conditions
* Mentally handicapped patients
* Patients with severe neurological conditions
* Patients of a nursing institution or other institutionalized patients
* Ward of the state / prisoner

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-11; Primary Completion 2020-12 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Rate of return of spontaneous circulation (ROSC) | 2-48h

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Schober, MD, Principal Investigator — Medical University Vienna, Austria, Dept. of Emergency Medicine
Locations (1):
- Medical University Vienna, Dept. of Emergency Medicine, Vienna, Austria